CLINICAL TRIAL: NCT00536926
Title: Telecommunication Via Cell Phones During Post-Operative Treatment After Lung Transplantation - an Open, Randomised Trial
Brief Title: Telecommunication Via Cell Phones During Post-Operative Treatment After Lung Transplantation
Acronym: TeleTx
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: Corscience, Inc. (Industry)
Responsible Party: Jens Gottlieb, M.D., Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 124
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2008-10

CONDITIONS: Lung Transplantation
Keywords: telemedicine; lung transplantation; home spirometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): home spirometry alone
  Interventions: Device: Home spirometer w/o BT
- B (Experimental): Home spirometry with data transfer via cellphone to clinical database
  Interventions: Device: Home spirometry with data transfer via cell phone; Device: Home spirometer with BT-cellphone

INTERVENTIONS:
Device: Home spirometry with data transfer via cell phone — home spirometry recording
  Other Names: Viasys AM1 /group A; Viasys AM1+BT/ group B
  Arms: B
Device: Home spirometer with BT-cellphone — Data transfer of home spirometry recordings via bluetooth to clinical database.
  Other Names: Viasys AM1 BT (Jaeger, Germany) with BT-cellphone
  Arms: B
Device: Home spirometer w/o BT — Standard home spirometry
  Other Names: Viasys (Jaeger, Germany) AM1
  Arms: A

SUMMARY:
In an investigation should be evaluated in contrast to a control group with standard post-treatment therapy (using home spirometry) after lung transplantation if transfer of home spirometry recordings to the transplant center via cell phones will lead to less complications, cost savings and bigger constancy of therapy.

DETAILED DESCRIPTION:
Home spirometry is used as a standard of care in lung transplant recipients in many centers worldwide. In case of deteriorating lung function response until therapy depends on patients efforts to reach the transplant center and the contactability of the transplant center.

Therefore transfer of home spirometry recordings to the transplant center via cell phones will lead to less complications, cost savings and bigger constancy of therapy compared to the home spirometry alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients after lung transplantation (single and double lung transplantation incl. combined organ transplantation) before hospital discharge

Exclusion Criteria:

* Dependency on long term care
* Restricted ability to communicate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-07; Primary Completion 2008-11 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Adherence | 6 months

SECONDARY OUTCOMES:
Latency: symptom onset to transplant team contact patient contacts emergency visits hospitalisations | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jens Gottlieb, MD, Principal Investigator — Dpt. Respiratory Medicine
Locations (1):
- Hannover Medical School, Dpt. resiratory Medicine OE6870, Hanover, Germany

REFERENCES:
- [Result] Sengpiel J, Fuehner T, Kugler C, Avsar M, Bodmann I, Boemke A, Simon A, Welte T, Gottlieb J. Use of telehealth technology for home spirometry after lung transplantation: a randomized controlled trial. Prog Transplant. 2010 Dec;20(4):310-7. doi: 10.1177/152692481002000402. PMID 21265282